CLINICAL TRIAL: NCT06671405
Title: An Open-label Study in Healthy Participants to Assess the Pharmacokinetics of AZD0780 When Administered Alone and in Combination With Itraconazole or Carbamazepine, and to Assess the Pharmacokinetics of Midazolam, and Ethinyl Estradiol/Levonorgestrel When Administered Alone and in Combination With AZD0780
Brief Title: An Open-label Study in Healthy Participants to Evaluate AZD0780 as an Object or Precipitant of CYP3A4-mediated Drug-drug Interactions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: D7960C00011
Record Dates: First submitted 2024-09-23; First posted 2024-11-04 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Dyslipidaemia
MeSH Terms: conditions — Dyslipidemias | interventions — Itraconazole; Carbamazepine; Midazolam; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Intervention Model Description: DDI study, open label, fixed sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Itraconazole Cohort (Experimental): * All participants will receive 2 single doses of dose 1 of AZD0780 and 14 doses of itraconazole, under fed conditions.
  * This part will consist of Period 1 (AZD0780 administration only), Period 2 (itraconazole administration only), and Period 3 (AZD0780 + itraconazole administration).
  Interventions: Drug: AZD0780; Drug: Itraconazole
- Carbamazepine Cohort (Experimental): * All participants will receive 2 single doses of dose 1 of AZD0780 and 6 doses of 100 mg, 6 doses of 200 mg, and 40 doses of 300 mg carbamazepine, under fed conditions.
  * This part will consist of Period 1 (AZD0780 administration only), Period 2 (carbamazepine administration only), and Period 3 (AZD0780 + carbamazepine administration)
  Interventions: Drug: AZD0780; Drug: Carbamazepine
- Midazolam Cohort (Experimental): * All participants will receive 10 single doses of AZD0780 dose 2 and 2 doses of midazolam. On midazolam dosing days, participants will receive midazolam under fasted conditions.
  * This part will consist of Period 1 (midazolam administration only), Period 2 (AZD0780 administration only), and Period 3 (AZD0780 + midazolam administration).
  Interventions: Drug: AZD0780; Drug: Midazolam
- EE and LNG Cohort (Experimental): * All participants will receive 15 single doses of AZD0780 dose 2 and 2 doses of EE and LNG. On EE and LNG dosing days, participants will receive EE and LNG under fasted conditions.
  * This part will consist of Period 1 (EE and LNG administration only), Period 2 (AZD0780 administration only), and Period 3 (AZD0780 + EE and LNG administration).
  Interventions: Drug: AZD0780; Drug: Ethinyl estradiol/levonorgestrel

INTERVENTIONS:
Drug: AZD0780 — Dose 1 and Dose 2
Drug: Itraconazole — * Period 2 (itraconazole administration only).
  * Period 3 (AZD0780 + itraconazole administration).
  Arms: Itraconazole Cohort
Drug: Carbamazepine — * Period 2 (carbamazepine administration only).
  * Period 3 (AZD0780 + carbamazepine administration only).
  Arms: Carbamazepine Cohort
Drug: Midazolam — * Period 1 (midazolam administration only).
  * Period 3 (AZD0780 + midazolam administration).
  Arms: Midazolam Cohort
Drug: Ethinyl estradiol/levonorgestrel — * Period 1 (EE and LNG administration only).
  * Period 3 (AZD0780 + EE and LNG administration).
  Arms: EE and LNG Cohort

SUMMARY:
An open-label, fixed sequence study in healthy participants to assess the pharmacokinetics of AZD0780 when administered alone and in combination with itraconazole and carbamazepine, and to assess the pharmacokinetics of midazolam and ethinyl estradiol/levonorgestrel (EE and LNG) when administered alone and in combination with AZD0780.

DETAILED DESCRIPTION:
The purpose of this study is to quantify the effect of itraconazole, a strong CYP3A inhibitor, and carbamazepine, a strong CYP3A inducer, on the PK of AZD0780 in healthy participants. This study will also evaluate AZD0780 as a precipitant of CYP3A4 mediated DDI by examining the PK of midazolam (a CYP3A4 substrate) and EE and LNG (CYP3A4 substrates) alone and in combination with AZD0780 in healthy participants.

The study duration (including screening period) will be approximately 9 to 10 weeks for Part 1, 12 to 14 weeks for Part 2, 6 to 8 weeks for Part 3, and 8 to 10 weeks for Part 4 (optional).

Study visits and treatment:

* Part 1: Participants who are eligible to participate in this study will stay at the Clinical Unit from Day -1 to Day 24 and return to the Clinical Unit again for a Follow-up Visit, 7 to 14 days after the last PK sample.
* Part 2: Participants who are eligible to participate in this study will stay at the Clinical Unit from Day -1 to Day 37 and return to the Clinical Unit again for a Follow-up Visit, 7 to 14 days after the last PK sample.
* Part 3: Participants who are eligible to participate in this study will stay at the Clinical Unit from Day -1 to Day 12 and return to the Clinical Unit again for a Follow-up Visit, 7 to 14 days after the last PK sample.
* Part 4 (optional): Participants who are eligible to participate in this study will stay at the Clinical Unit from Day -1 to Day 22 and return to the Clinical Unit again for a Follow-up Visit, 7 to 14 days after the last PK sample.

Number of Participants:

Approximately 78 participants will be enrolled in this study; 18 participants in Part 1 (itraconazole Cohort), 24 participants in Part 2 (carbamazepine Cohort), 18 participants in Part 3 (midazolam Cohort), and 18 Participants in Part 4 (EE and LNG Cohort) (optional).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study-specific procedures.
2. Healthy male and female participants of non-childbearing potential aged 18 to 75 years with suitable veins for cannulation or repeated venipuncture. Part 4 only: Healthy female participants of non-childbearing potential aged 18 to 75 years with suitable veins for cannulation or repeated venipuncture.
3. All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
4. Females of non-childbearing potential must be confirmed at the Screening Visit by fulfilling one of the following criteria:

   1. Postmenopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and FSH levels in the postmenopausal range.
   2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation or tubal occlusion.
5. Sexually active fertile male participants with partners of childbearing potential must adhere to the contraception methods detailed in Appendix C 2.1 from the time of first administration of AZD0780 administration until 3 months after the study Follow-up Visit.
6. Have a BMI between 18 and 35 kg/m2 inclusive and weight at least 50 kg at the Screening Visit and on admission to the Clinical Unit.

Exclusion Criteria:

1. History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any prior gastrointestinal surgery which may affect absorption, eg, gastric bypass or resection.
4. Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
5. Any laboratory values with the following deviations at the Screening Visit or on admission to the Clinical Unit. Abnormal values may be repeated once at the discretion of the Investigator.
6. Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis results other than those described under exclusion criterion number 5, at screening and/or admission to the Clinical Unit, as judged by the Investigator. Abnormal values may be repeated once at the discretion of the Investigator.
7. Any positive result at Screening for serum HBsAg, HBcAb, HCV, or HIV.
8. Any clinically significant abnormal findings in abnormal vital signs, after at least 10 minutes supine rest, at Screening and on admission to the Clinical Unit, as judged by the Investigator. Abnormal values may be repeated once at the discretion of the Investigator..
9. Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG as considered by the Investigator that may interfere with the interpretation of QTc interval changes.
10. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 3 months prior to screening.
11. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the Investigator.
12. Positive screen for drugs of abuse, alcohol, or cotinine at Screening or on admission to the Clinical Unit.
13. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD0780, itraconazole (Part 1 only), carbamazepine (Part 2 only), midazolam (Part 3 only), or EE/LNG (Part 4 only).
14. Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) defined as the regular consumption of more than 500 mg of caffeine per day (eg, > 5 cups of coffee [one cup ~100 mg caffeine]; one cup of tea ~30 mg caffeine) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the Clinical Unit.
15. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of study intervention.
16. Use of any prescribed or nonprescribed medication including hormone replacement therapy, antacids or acid reducing agents (including proton pump inhibitors),analgesics (other than paracetamol/acetaminophen), herbal remedies, mega dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of study intervention or longer if the medication has a long half-life.
17. Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
18. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days or 5 half-lives (whichever is longest) of the first administration of the study intervention in this study. NOTE: participants consented and screened, but not enrolled/randomized in this study or a previous Phase I study, are not excluded. NOTE: All follow-up activities in a previous research study (including last study visit, unresolved AEs, or abnormal laboratory values) have to be completed prior to the Screening Visit. NOTE: Participants must be checked in VCT in the USA.
19. Participants who have previously received AZD0780 within 60 days prior to Screening.
20. Current/previous use of drugs that reduce or inhibit PCSK9 (approved or investigational; within 12 months of enrolment). Any current/previous use of inclisiran.
21. Elevated or abnormal liver enzymes or active liver disease, or who have experienced liver toxicity with other drugs.
22. Known or confirmed for HLA-A*3101 and/or HLA-B*1502 allele at Screening (Part 2 only).
23. Participant who previously experienced hypersensitivity reaction to anticonvulsants including phenytoin, primidone, and phenobarbital.
24. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the Clinical Unit).
25. Judgment by the Investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the Screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
26. Participants who are vegans or have medical dietary restrictions.
27. Participants who cannot communicate reliably with the Investigator.
28. Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
AUCinf (Area under concentration-time curve from time 0 to infinity) | Period 1 (Day 1 to 11 Cohort 1 and Cohort 2) and Period 3 (Day 14-24 Part 1 and Day 27-37 Part 2)
  To describe the PK of AZD0780 when administered alone and in combination with itraconazole and carbamazepine.
AUClast (Area under concentration curve from time 0 to the last quantifiable concentration) | Period 1 (Day 1 to 11 Cohort 1 and Cohort 2) and Period 3 (Day 14-24 Part 1 and Day 27-37 Part 2)
  To describe the PK of AZD0780 when administered alone and in combination with itraconazole and carbamazepine.
Cmax (Maximum observed drug concentration) | Period 1 (Day 1 to 11 Cohort 1 and Cohort 2) and Period 3 (Day 14-24 Part 1 and Day 27-37 Part 2)
  To describe the PK of AZD0780 when administered alone and in combination with itraconazole and carbamazepine.
AUCinf | Period 1 (Day 1 to 2 Part 3 and Day 1 to 7 Part 4) and Period 3 (Day 11-12 Part 3 and Day 16 to 22 Part 4)
  To assess the effect of AZD0780 on the PK of midazolam (Part 3) and EE and LNG (Part 4).
AUClast | Period 1 (Day 1 to 2 Part 3 and Day 1 to 7 Part 4) and Period 3 (Day 11-12 Part 3 and Day 16 to 22 Part 4)
  To assess the effect of AZD0780 on the PK of midazolam (Part 3) and EE and LNG (Part 4).
Cmax | Period 1 (Day 1 to 2 Part 3 and Day 1 to 7 Part 4) and Period 3 (Day 11-12 Part 3 and Day 16 to 22 Part 4)
  To assess the effect of AZD0780 on the PK of midazolam (Part 3) and EE and LNG (Part 4).

SECONDARY OUTCOMES:
CL/F (Apparent total body clearance) | Period 1 (Day 1 to 11 Cohort 1 and Cohort 2) and Period 3 (Day 14-24 Part 1 and Day 27-37 Part 2)
  To describe the PK of AZD0780 when administered alone, in combination with itraconazole or in combination with carbamazepine.
t½λz (Terminal elimination half-life) | Period 1 (Day 1 to 11 Cohort 1 and Cohort 2) and Period 3 (Day 14-24 Part 1 and Day 27-37 Part 2)
  To describe the PK of AZD0780 when administered alone, in combination with itraconazole or in combination with carbamazepine.
tmax (Time to reach maximum observed concentration) | Period 1 (Day 1 to 11 Cohort 1 and Cohort 2) and Period 3 (Day 14-24 Part 1 and Day 27-37 Part 2)
  To describe the PK of AZD0780 when administered alone, in combination with itraconazole or in combination with carbamazepine.
Vz/F (Apparent volume of distribution based on the terminal phase) | Period 1 (Day 1 to 11 Cohort 1 and Cohort 2) and Period 3 (Day 14-24 Part 1 and Day 27-37 Part 2)
  To describe the PK of AZD0780 when administered alone, in combination with itraconazole or in combination with carbamazepine.
Number of participants with Adverse Events and Serious Adverse Events (AEs and SAEs) | From Baseline until Follow-up Visit (7 to 14 days post-discharge)
  To assess the safety and tolerability of AZD0780 when administered alone and in combination with itraconazole, carbamazepine, midazolam and EE and LNG.
Number of participants with treatment emergent abnormal ECGs | From Baseline until Follow-up Visit (7 to 14 days post-discharge)
  To assess the safety and tolerability of AZD0780 when administered alone and in combination with itraconazole, carbamazepine, midazolam and EE and LNG.
Vital signs and laboratory test results | From Baseline until Follow-up Visit (7 to 14 days post-discharge)
  To assess the safety and tolerability of AZD0780 when administered alone and in combination with itraconazole, carbamazepine, midazolam and EE and LNG.
CL/F | Period 1 (Day 1 to 2 Part 3 and Day 1 to 7 Part 4) and Period 3 (Day 11-12 Part 3 and Day 16 to 22 Part 4)
  To describe the PK of midazolam (Part 3) and EE and LNG (Part 4) when administered alone and in combination with AZD0780.
t½λz | Period 1 (Day 1 to 2 Part 3 and Day 1 to 7 Part 4) and Period 3 (Day 11-12 Part 3 and Day 16 to 22 Part 4)
  To describe the PK of midazolam (Part 3) and EE and LNG (Part 4) when administered alone and in combination with AZD0780.
tmax | Period 1 (Day 1 to 2 Part 3 and Day 1 to 7 Part 4) and Period 3 (Day 11-12 Part 3 and Day 16 to 22 Part 4)
  TTo describe the PK of midazolam (Part 3) and EE and LNG (Part 4) when administered alone and in combination with AZD0780.
Vz/F | Period 1 (Day 1 to 2 Part 3 and Day 1 to 7 Part 4) and Period 3 (Day 11-12 Part 3 and Day 16 to 22 Part 4)
  To describe the PK of midazolam (Part 3) and EE and LNG (Part 4) when administered alone and in combination with AZD0780.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States